CLINICAL TRIAL: NCT04599842
Title: Analgesic Effect of Erector Spinae Plane Block After Caesarean Section: A Randomized Controlled Trial
Brief Title: Analgesic Effect of Erector Spinae Plane Block After Caesarean Section
Acronym: AnESPaCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, MD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/1
Record Dates: First submitted 2020-10-09; First posted 2020-10-23 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Ceserean Section and Postoperative Pain
Keywords: Ceserean section, ESP block, postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP SA (No Intervention): Group SA was categorized as the group which spinal anaesthesia alone (SA) was performed
- GROUP SA+ESP (Active Comparator): Group SA+ESP was categorized as group which SA+ESP block was performed.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector Spinae Plane block is performed by giving local anesthetic to the plan between the erector spinae muscle and the transverse process.
  Arms: GROUP SA+ESP

SUMMARY:
Background: Our hypothesis was that bilateral ESP block applied from the transverse process of T9 in women who underwent elective cesarean section with pfannenstiel incision under spinal anesthesia could provide effective postoperative analgesia.The primary outcome in this study was total opioid consumption for 24 hours.

Material and Method: This randomized prospective study was carried out on 50 pregnant women who was scheduled for elective cesarean delivery via a Pfannenstiel incision with spinal anesthesia.Patients were randomly allocated in to two equal groups.Group SA was categorized as the group which spinal anaesthesia alone (SA) was performed, Group SA+ESP was categorized as group which SA+ESP block was performed. All groups received 7 mg isobaric bupivacaine +15 µg fentanyl intrathecally through spinal anesthesia. The SA+ESP group, ESP block was performed at the ninth thoracic transverse process with 20 ml 0.25% bupivacaine + 2 mg dexamethasone immediately after the operation. Total fentanyl consumption in 24 hrs, visual analogue scale (VAS) score for pain, time to the first analgesic request were evaluated postoperatively.

ELIGIBILITY:
Inclusion Criteria:pregnant women,38-42 gestational weeks, ASA I-II

Exclusion Criteria:

* ≤18 or ≥45 age, has emergency obstetric surgery, pregnancy induced hypertension, significantly systematic disease, foetal or placental abnormality, hypersensitivity or allergy history to medicine to be used in the study, BMI≥35, autonomic neuropathy, diabetic, contraindicate to apply neuroachylic anaesthesia, who was transferred to general anaesthesia, could not decide or did not want to participate in the study, had severe respiratory and cardiac disease, was transferred to general anaesthesia, has infection, spine or chest wall deformity in operation area, has opioid dependence, chronic analgesic usage, inability to use a patient-controlled analgesia (PCA) device, couldn't be able to cooperative and express their pain with visual analogue scale score (VAS).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 50 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
The primary outcome in this study was total opioid consumption for 24 hours. | 24 hours
  Total fentanyl consumption postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Ince, MD, Study Director — Ataturk University, Department of Anesthesiology and Reanimation
Locations (1):
- Aysenur Dostbil, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided